CLINICAL TRIAL: NCT07405593
Title: The Combination Model of 30 Degree Head Up and Murottal Therapy on Blood Pressure, Pulse Rate, Respiratory Rate, Pain Degree, and Projectile Vomiting in Stroke Patients
Brief Title: Head Up Position and Murottal Therapy in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fila Diana Nurhayati, Graduate Researcher, Universitas Muhammadiyah Surakarta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FDN-HU-MUROTTAL-STROKE-2026
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Head Up; Murottal Therapy
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are assigned in parallel to an intervention group receiving 30-degree head-up positioning and murottal therapy or to a control group receiving standard care.
Masking Description: This study is conducted as an open-label trial because the non-pharmacological interventions, including 30-degree head-up positioning and murottal therapy, are clearly observable and cannot be feasibly blinded to participants, care providers, or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of 30-Degree Head-Up Positioning and Murottal Therapy (Experimental): Participants receive a combination of 30-degree head-up positioning and murottal therapy in addition to standard nursing care during the intervention period.
  Interventions: Other: Combination of 30 Degree Head Up and Murottal Therapy
- Standard Care (Active Comparator): Participants receive standard nursing care according to the hospital's clinical protocol without the addition of head-up positioning or murottal therapy.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Combination of 30 Degree Head Up and Murottal Therapy — Participants in this group received a combination of two non-pharmacological interventions during the study period. First, participants were positioned with their heads elevated at a 30-degree angle while lying in bed to support physiological stability, including monitoring of blood pressure, pulse rate, respiratory rate, pain level, and projectile vomiting. Second, participants listened to Quranic recitation (murottal therapy) via audio recording in a quiet environment. Both interventions were administered simultaneously. Intervention sessions lasted 30 minutes for 3 days (a consistent duration and frequency for all participants in this group). Outcomes such as vital signs, pain level, and episodes of severe vomiting were monitored before and after the intervention period.
  Arms: Combination of 30-Degree Head-Up Positioning and Murottal Therapy
Other: Standard Care (in control arm) — Participants in this arm receive standard nursing care according to the hospital protocol without additional head-up positioning or murottal therapy. Standard care includes routine monitoring of vital signs, medication administration, and basic supportive nursing interventions.
  Arms: Standard Care

SUMMARY:
This study aims to evaluate the effects of a combination of a 30-degree head-up position and murottal therapy on physiological and symptom outcomes in stroke patients. The intervention is expected to influence blood pressure, pulse rate, respiratory rate, pain level, and the incidence of projectile vomiting. Stroke patients will receive standard care with the addition of the combined intervention. The results of this study may support non-pharmacological nursing interventions to improve patient comfort and clinical stability.

DETAILED DESCRIPTION:
Stroke patients often experience physiological instability and discomfort, including changes in blood pressure, pulse rate, respiratory rate, pain, and nausea or vomiting. Non-pharmacological nursing interventions are needed to support patient comfort and clinical stability during acute care. Head-up positioning and murottal therapy are commonly used supportive interventions in nursing practice, but evidence regarding their combined effects remains limited.

This study aims to evaluate the effects of a combination of a 30-degree head-up position and murottal therapy on blood pressure, pulse rate, respiratory rate, pain degree, and projectile vomiting in stroke patients. The study involves stroke patients receiving standard medical and nursing care, with the addition of the combined intervention as part of supportive nursing management.

The head-up position will be applied at a 30-degree angle, while murottal therapy will be delivered through 30-minute audio recitation during for 3 days. Physiological parameters and symptom outcomes will be measured before and after the intervention according to the study protocol. The findings of this study are expected to contribute evidence for the use of simple, non-pharmacological nursing interventions to improve comfort and physiological responses in stroke patients.

ELIGIBILITY:
Inclusion Criteria :

1. Patients with a medical diagnosis of stroke (hemorrhagic and non-hemorrhagic).
2. Patients with systolic blood pressure above 150 mmHg.
3. Somnolence (GCS ≥ 9).
4. Muslim.
5. Patients without hearing impairment.
6. Willingness to participate and sign informed consent.

Exclusion criteria :

1. Patients who are non-Muslim.
2. Patients with decreased consciousness (GCS < 9).
3. Patients with heart problems.
4. Patients with psychiatric disorders.
5. Patients receiving sedative therapy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline and after completion of the 3-day intervention
  Change in systolic and diastolic blood pressure from baseline to after completion of the 3-day intervention.
Pulse Rate | Baseline and after completion of the 3-day intervention
  Change in pulse rate from baseline to after completion of the 3-day intervention.
Respiratory Rate | Baseline and after completion of the 3-day intervention
  Change in respiratory rate from baseline to after completion of the 3-day intervention
Pain Degree | Baseline and after completion of the 3-day intervention
  Change in pain score measured using the Critical-Care Pain Observation Tool (CPOT; range 0-8), where higher scores indicate more severe pain, from baseline to after completion of the 3-day intervention.
Projectile Vomiting | Baseline and after completion of the 3-day intervention
  Change in nausea and vomiting severity measured using the Rhodes Index of Nausea, Vomiting, and Retching (RINVR; range 0-32), where higher scores indicate more severe symptoms, from baseline to after completion of the 3-day intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Indriati Solo Baru, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Intracranial Pressure Monitoring and Management in Aneurysmal Subarachnoid Hemorrhage — https://doi.org/10.1007/s12028-023-01752-y
- See also: Adherence to Head-of-Bed Elevation in Traumatic Brain Injury: An Audit. — https://doi.org/10.1055/s-0042-1758749
- See also: Interdisciplinary Neurosurgery : Advanced Techniques and Case Management Position-dependent hemodynamic changes in neurosurgery patients : A narrative review. — https://doi.org/10.1016/j.inat.2023.101886
- See also: Nausea and vomiting in pregnancy ( NVP ) in Chinese pregnant women : a cross-sectional study — https://doi.org/10.1186/s12884-024-06686-7
- See also: Associations between computed tomography markers of cerebral small vessel disease and hemorrhagic transformation after intravenous thrombolysis in acute ischemic stroke patients. — https://doi.org/10.3389/fneur.2023.1144564
- See also: Blood Pressure Management Pre- and Post-Reperfusion in Acute Ischemic Stroke: Evidence and Insights from Recent Studies. — https://doi.org/10.1007/s11910-025-01443-5
- See also: Measuring pain intensity in older patients : a comparison of five scales. — https://doi.org/10.1186/s12877-024-05127-6
- See also: The Impact of Listening to , Reciting , or Memorizing the Quran on Physical and Mental Health of Muslims : Evidence From Systematic Review — https://doi.org/10.3389/ijph.2022.1604998